CLINICAL TRIAL: NCT06214182
Title: A Study of Immune Heterogeneity Before and After Cardiopulmonary Bypass in Children Undergoing Cardiac Surgery Based on ScRNA-seq
Brief Title: Immune Heterogeneity Before and After Cardiopulmonary Bypass in Children
Status: Completed | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Wenyuan Zhang, Principal Investigator, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2023-IRB-0303-P-01
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group T1: T1 is before CPB.
- Group T2: T2 is 2 hours after CPB.
- Group T3: T3 is 3 days after CPB.

SUMMARY:
The goal of this observational study is to learn about functional heterogeneity of immune cells before and after cardiopulmonary bypass (CPB) in children with congenital heart disease (CHD). The main question[s] it aims to answer are:

* Does CPB cause immune paralysis after CHD surgery?
* How does the functional heterogeneity of immune cells change before and after CPB in children undergoing CHD surgery? Participants will receive 3ml of peripheral blood before CPB, 2 hours after CPB, and 3 days after CPB, and the peripheral blood samples will be sequenced by single cell to explore the immune heterogeneity before and after CPB.

DETAILED DESCRIPTION:
CPB-induced immune paralysis is the main cause of postoperative infection in CHD, which seriously affects the prognosis of children. The underlying mechanism of CPB-induced immune paralysis has not been fully determined. This study intends to use scRNA-seq to describe gene transcription profiles of immune cells in peripheral blood of children undergoing CHD surgery before and after CPB, and explore the differences within and between different immune cell populations including T cells and the changes of immune cells in different sequences. To fill the gap in the study of immune mechanism in CPB-induced immune paralysis microenvironment at single-cell resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight range: 2500-6000g;
2. Operation duration >90min;

Exclusion Criteria:

1. preterm infants or preoperative infections;
2. systemic immune diseases and serious complications: such as rheumatoid arthritis, systemic lupus erythematosus, severe liver and kidney function damage, leukemia, etc.;
3. Patients who have received an organ transplant;
4. Patients who have received immunomodulatory drugs: patients who have received immunomodulatory drugs before surgery;
5. Parents refused to participate or were unable to provide sufficient samples: Parents or legal guardians refused to participate in the study.

Ages: 31 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In this study, children aged 31d-1y who underwent subCPB ventricular septal defect repair for the first time between January 2024 and February 2024 at the Children's Hospital Affiliated to Zhejiang University School of Medicine were enrolled. This study will comply with the requirements set out in the Declaration of Helsinki and will be approved by the Ethics Committee of our Institute.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Expression of genes | From enrollment to the end of CPB at 3 days
  The gene expression in single cells of peripheral blood samples was detected

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided